CLINICAL TRIAL: NCT06309511
Title: Subendocardial Viability Ratio in Hypertension
Acronym: SEVR-HT
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C218
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
Keywords: Myocardial ischemia; Buckberg index
MeSH Terms: conditions — Hypertension; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Arterial tonometry — Arterial transcutaneous tonometry

SUMMARY:
The aim of the research is to evaluate the Subendocardial Viability Ratio (SEVR) in hypertensive patients, using non-invasive arterial tonometry, and to establish the influencing factors and the possibility of predicting cardiovascular morbidity and mortality in arterial hypertension.

The SEVR will be evaluated on all patients belonging to the Arterial Hypertension Centers undergoing non-invasive arterial tonometry.

The SEVR is calculated on the morphology of the central pressure wave as the ratio between the DPTI (diastolic pressure-time index), i.e. the area between the carotid pressure curve and the ventricular pressure curve during the diastolic phase, and the SPTI ( systolic pressure-time index), i.e. the area under the carotid pressure curve during the systolic phase.

The SEVR will be correlated with the anthropometric and pathology variables which will be collected in an appropriate database.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension

Exclusion Criteria:

* Atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Buckberg index | At recruitment, at 1 year, 2 years, 3 years and 4 years of follow-up
  Assessment of subendocardial viability ratio (SEVR)

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Centro di Prevenzione e Cura dell'Ipertensione Arteriosa "Alessandro Filippi", Mascalucia, Catania
  - Unità Operativa Semplice Dipartimentale Ipertensione Arteriosa "Anna Maria Pirrelli", Università degli Studi di Bari "Aldo Moro". Policlinico Consorziale di Bari, Bari
  - Istituto Auxologico Italiano IRCCS, Milan
  - Medicina II Cardiovascolare, AUSL-IRCCS di Reggio Emilia, Reggio Emilia
  - Dipartimento di Scienze Mediche, Chirurgiche e della Salute, Università degli studi di Trieste, Trieste

IPD SHARING:
Plan to Share IPD: No